CLINICAL TRIAL: NCT00601042
Title: Randomized, Placebo-controlled, Double-blind, Phase IV Trial to Assess the Efficacy of a Traditional Swedish Smokeless Tobacco Product ("Snus") to Reduce or Replace Cigarette Smoking Among Adult Smokers in Serbia
Brief Title: Serbian Smoking Reduction/Cessation Trial (2SRT)
Acronym: 2SRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Match AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 07-01; SM 07-01
Record Dates: First submitted 2007-12-27; First posted 2008-01-25 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Cigarette Smoking
Keywords: smoking reduction; smoking cessation; randomized trial; Swedish snus; smokeless tobacco
MeSH Terms: conditions — Cigarette Smoking; Smoking Reduction; Smoking Cessation; Tobacco Use | interventions — Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Swedish snus ad libitum as a substitute for cigarettes
  Interventions: Other: Swedish snus (smokeless tobacco)
- 2 (Placebo Comparator): Tobacco-free, nicotine-free placebo snus ad libitum as a substitute for cigarettes
  Interventions: Other: Onico

INTERVENTIONS:
Other: Swedish snus (smokeless tobacco) — Snus in sachets 1.0 g or 0.5 g, 2 flavors. Usage ad libitum.
  Arms: 1
Other: Onico — Tobacco-free, nicotine-free placebo snus, 2 sachet sizes (1.0 g, 0.5 g), 2 flavors (same as in the experimental arm). Usage ad libitum.
  Other Names: Onico (brand name)
  Arms: 2

SUMMARY:
The study aims to establish if a low-nitrosamine, smokeless tobacco product (Swedish snus) can help adult smokers to reduce and eventually completely quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Male and female smokers in good general health aged 20-65 years regularly smoking >10 cigarettes per day for more than 1 year who are motivated to reduce or quit smoking

Exclusion Criteria:

* Subjects with uncontrolled hypertension, history of coronary heart disease or other significant heart condition
* History of other significant medical condition that might interfere with study procedures
* Pregnant or nursing mother
* Current drug abuse.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Smoking reduction defined as a reduction in self-reported number of smoked cigarettes per day >50% compared to base-line, verified by a reduction in CO in exhaled air of >1 ppm compared to base-line | 6 months

SECONDARY OUTCOMES:
Smoking cessation defined as self-reported total abstention from cigarettes verified by CO in exhaled air <10 ppm | 3, 6, 9 and 12 months
Clinical tests and biomarkers relevant for exposure to tobacco | 3, 6, 9, and 12 months
Smoking reduction | 12, 24, 36 and 48 months
  Smoking reduction according to self-report
Smoking reduction | 12, 24, 36 and 48 months
  Smoking reduction compared to baseline according to self-report

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Joksic, Ph D, Principal Investigator — Institute for Nuclear Research "Vinca", Belgrade, Serbia; Robert Nilsson, Ph D, Prof, Study Chair — Stockholm University, Stockholm, Sweden
Locations (2):
- Serbia (2):
  - Institute of Nuclear Sciences "Vinca", Belgrade
  - Ambulanta Medicine Rada, Nis-Jugopetrol, New Belgrade

REFERENCES:
- [Result] Joksic G, Spasojevic-Tisma V, Antic R, Nilsson R, Rutqvist LE. Randomized, placebo-controlled, double-blind trial of Swedish snus for smoking reduction and cessation. Harm Reduct J. 2011 Sep 13;8:25. doi: 10.1186/1477-7517-8-25. PMID 21914165